CLINICAL TRIAL: NCT02968641
Title: A Phase 2b, Open-Label, Randomized Study of the Safety, Tolerability, and Pharmacodynamic Activity of Lonafarnib With or Without Ritonavir in Patients Chronically Infected With Hepatitis Delta Virus (LOWR-5)
Brief Title: A Study of Lonafarnib With or Without Ritonavir in Patients With HDV
Acronym: LOWR-5
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was initially planned to enroll patients in Mongolia. However, due to challenges in setting it up in Mongolia, this study was later determined not to be initiated.
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIG-LNF-004
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Chronic Delta Hepatitis
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — lonafarnib; Ritonavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LNF 25 mg bid and RTV 100 mg bid (Active Comparator): Patients will take lonafarnib 25 mg BID and ritonavir 100 mg BID. Patients will also take an anti-hepatitis B virus (HBV) nucleos(t)ide analog (NUC) from the first dose of LNF through the end of the study.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir
- LNF 50 mg bid and RTV 100 mg bid (Active Comparator): Patients will take lonafarnib 50 mg BID and ritonavir 100 mg BID. Patients will also take an anti-hepatitis B virus (HBV) nucleos(t)ide analog (NUC) from the first dose of LNF through the end of the study.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir
- LNF 100 mg bid (Active Comparator): Patients will take lonafarnib 100 mg BID. Patients will also take an anti-hepatitis B virus (HBV) nucleos(t)ide analog (NUC) from the first dose of LNF through the end of the study.
  Interventions: Drug: Lonafarnib

INTERVENTIONS:
Drug: Lonafarnib — antiviral farnesyltransferase inhibitor
  Other Names: EBP994; Sarasar
Drug: Ritonavir — CYP 3A4 inhibitor, lonafarnib booster
  Other Names: Norvir
  Arms: LNF 25 mg bid and RTV 100 mg bid; LNF 50 mg bid and RTV 100 mg bid

SUMMARY:
A Phase 2b, Open-Label, Randomized Study of the Safety, Tolerability, and Pharmacodynamic Activity of Lonafarnib With or Without Ritonavir in Patients Chronically Infected with Hepatitis Delta Virus

DETAILED DESCRIPTION:
This Phase 2b, randomized, open-label study will assess the safety, tolerability, and pharmacodynamics (PD)/efficacy of 48 weeks of lonafarnib (LNF) and ritonavir (RTV) combination therapy vs. LNF monotherapy in patients with chronically infected with Hepatitis Delta Virus (CHD). Sixty patients will be enrolled at a single study site. Eligible patients will have CHD infection (≥ 6 months) confirmed by positive HDV antibody (Ab) test and HDV RNA ≥ 3 lg IU/mL by quantitative polymerase chain reaction (qPCR) at study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to comply with study procedures and provide written consent
2. 18 - 65 years old
3. Body mass index (BMI) of ≥ 18 kg/m2 and weighs ≥ 45 kg
4. CHD infection of at least 6 months' duration documented by a positive HDV antibody (Ab) test and HDV RNA ≥ 3 log10/mL by qPCR at study entry
5. Serum ALT > upper limit of the normal range (ULN) and < 10 × ULN
6. Liver biopsy within 12 months of Day 1 demonstrating evidence of chronic hepatitis. If no liver biopsy is available, the patient must be willing to consent to and have no contraindication to liver biopsy
7. ECGs demonstrating no acute ischemia or clinically significant abnormality and a QT interval corrected for heart rate (QTcF) < 450 ms for male patients and < 460 ms for female patients
8. Dilated retinal examination ≤ 1 year before screening: For patients with diabetes, hypertension, or other risk factors for retinal disease, performed by a licensed ocular specialist; for all other patients, a normal retinal examination as assessed by the investigator or a licensed ocular specialist
9. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use adequate methods of contraception during the study and for 90 days after the last dose of study drug. Female patients of childbearing potential are all those except patients who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal.

For females: 2 of the following contraceptive methods, with at least 1 being a barrier method:

* Hormonal contraceptives for ≥ 3 months before screening
* Intrauterine device (IUD) in place ≥ 3 months before screening
* Double-barrier methods (use of condom [male partner] with either diaphragm with spermicide or cervical cap with spermicide) from screening
* Surgical sterilization of the partner (vasectomy ≥ 1 month before screening)

For males:

* Surgical sterilization (vasectomy ≥ 1 month before screening) or
* Both of the following contraceptive methods from screening:

  * Consistently and correctly use a condom
  * Partner must agree to use a hormonal contraceptive or a nonhormonal barrier method (IUD or diaphragm with spermicide or cervical cap with spermicide)

Exclusion Criteria:

General Exclusions

1. Participation in a clinical trial with, or use of, any investigational agent within 30 days before screening
2. Previous use of LNF.
3. Female patients who are pregnant or breastfeeding. Male patients must confirm that their female sexual partners are not pregnant. Female patients must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of any investigational agent).

   Exclusions Based on Disease
4. Current or previous history of decompensated liver disease (Child-Pugh Class B or C)
5. Co-infected with human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
6. Positive results for HIV or HCV Ab at screening. Patients with a positive HCV Ab at screening are allowed if they have completed a curative antiviral regimen and have documented undetectable HCV RNA for at least 3 months before screening and at screening.
7. Past history or current evidence of decompensated liver disease, defined as any of the following at screening:

   * Bilirubin level ≥ 2.5 mg/dL unless due to Gilbert's disease
   * Serum albumin level < 3.0 g/dL
   * International normalized ratio (INR) ≥ 1.5
8. Evidence of significant portal hypertension such as hepatic venous pressure gradient (HVPG) ≥ 10 mmHg; current presence or history of esophageal or abdominal varices, variceal bleeding, or splenomegaly > 12 cm length on imaging
9. Current evidence or history of ascites requiring diuretics or paracentesis, or hepatic encephalopathy
10. Current evidence or history of hepatic encephalopathy
11. Any of the following abnormal laboratory test results at screening:

    * Platelet count < 90,000 cells/mm3
    * White blood cell (WBC) count < 3,000 cells/mm3
    * Absolute neutrophil count (ANC) < 1,500 cells/mm3
    * Hemoglobin

      * < 11 g/dL for women
      * < 12 g/dL for men
    * Serum creatinine concentration ≥ 1.5 × ULN
    * Confirmed creatinine clearance (CrCl) < 50 mL/min by Cockroft-Gault or an estimated glomerular filtration rate (eGFR) > 80 mL/min at screening, based on the Cockcroft-Gault equation
    * Alpha-fetoprotein ≥ 100 ng/mL
12. Evidence of another form of viral hepatitis or another form of liver disease (eg, autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, alcoholic liver disease, nonalcoholic steatohepatitis, hemochromatosis, alpha-1-anti-trypsin deficiency)
13. History of hepatocellular carcinoma
14. Patients with any of the following:

    * Current eating disorder or alcohol abuse
    * Excessive alcohol intake, defined as follows:

      * > 20 g/day for females (1.5 standard alcohol drinks) or
      * > 30 g/day for males (2.0 standard alcohol drinks).
      * A standard drink contains 14 g of alcohol: 360 mL of beer, 150 mL of wine, or 45 mL of spirits
    * In the opinion of the investigator, an alcohol use pattern that will interfere with study conduct
    * Drug abuse within the previous 6 months before screening, with the exception of cannabinoids and their derivatives
15. Prior history or current evidence of any of the following:

    * Immunologically mediated disease (eg, rheumatoid arthritis, inflammatory bowel disease, severe psoriasis, systemic lupus erythematosus) that requires more than intermittent nonsteroidal anti-inflammatory medications for management or that requires use of systemic corticosteroids in the 6 months before screening (inhaled asthma medications are allowed)
    * Retinal disorder or clinically relevant ophthalmic disorder
    * Any malignancy within 5 years before screening. Exceptions are superficial dermatologic malignancies (eg, squamous cell or basal cell skin cancer treated with curative intent), or successfully treated in-situ carcinoma of the cervix.
    * Cardiomyopathy or significant ischemic cardiac or cerebrovascular disease (including history of angina, myocardial infarction, or interventional procedure for coronary artery disease)
    * Chronic pulmonary disease (eg, chronic obstructive pulmonary disease) associated with functional impairment
    * Pancreatitis
    * Severe or uncontrolled psychiatric disorder (eg, depression, manic condition, psychosis, acute and/or chronic cognitive dysfunction, suicidal behavior, and relapse of substance abuse)
    * Bone marrow or solid organ transplantation
16. Other significant medical condition that may require intervention during the study. Patients with any serious condition that, in the opinion of the investigator, would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed. Patients for whom participation in the study would increase their risk.

    Exclusions Based on Concurrent Medication Use
17. Any prescription or herbal product that is not approved by the investigator
18. Therapy with an immunomodulatory agent, IFN-alfa (IFN alfa-2a or IFN alfa-2b, or pegylated IFN alfa-2a or alfa-2b), cytotoxic agent, or systemic corticosteroids within 12 months before screening and during the study
19. Use of heparin or warfarin during the study
20. Systemic antibiotics, antifungals, or antivirals for treatment of active infection other than HBV within 14 days before study randomization or during the study
21. Long-term treatment (> 2 weeks) before or during the study with agents that have a high risk for nephrotoxicity or hepatotoxicity unless it is approved by the medical monitor
22. Receipt of systemic immunosuppressive therapy within 3 months before screening or during the study
23. History or evidence for any intolerance or hypersensitivity to LNF, RTV, or other substances that are part of the study drug
24. Concomitant use of any of the following:

    * Medications or foods that are known moderate or strong inducers or inhibitors of CYP3A4
    * Drugs known to prolong the PR or QT interval unless otherwise described in this protocol
    * Statins, due to inhibition of mevalonate synthesis, which reduces protein prenylation
25. Concomitant use of medications contraindicated in the prescribing information for RTV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HDV viral load at Week 72 visit (end of follow-up) | 72 weeks
  HDV RNA viral load will be quantified with a real-time qPCR assay with a lower limit of quantification (LLOQ) of 14 IU/mL

SECONDARY OUTCOMES:
Change from baseline in HDV viral load at Week 48 visit (end of treatment, EOT) | 48 weeks
Proportion of patients with histological response | 72 weeks
  Histological response defined as an improvement in liver histology by at least 2 points in the Hepatitis Activity Score (HAI) with improvement or no worsening of the fibrosis score, at the EOT compared with baseline
Proportion of patients with sustained virologic response: HDV RNA below the LLOQ 12 weeks after EOT (48 weeks) | 60 weeks
Proportion of patients with sustained virologic response: HDV RNA below the LLOQ 24 weeks after EOT (48 weeks) | 72 weeks
Number of participants with treatment-emergent changes in clinical laboratory findings | 48 weeks
Number of participants with treatment-emergent / treatment-related adverse events (AE) and serious adverse events | 48 weeks
Number of participants with AE leading to early discontinuation of study treatment or dose reduction | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo B Martins, MD, DPhil, Study Director — Eiger BioPharmaceuticals

REFERENCES:
- [Background] Koh C, Canini L, Dahari H, Zhao X, Uprichard SL, Haynes-Williams V, Winters MA, Subramanya G, Cooper SL, Pinto P, Wolff EF, Bishop R, Ai Thanda Han M, Cotler SJ, Kleiner DE, Keskin O, Idilman R, Yurdaydin C, Glenn JS, Heller T. Oral prenylation inhibition with lonafarnib in chronic hepatitis D infection: a proof-of-concept randomised, double-blind, placebo-controlled phase 2A trial. Lancet Infect Dis. 2015 Oct;15(10):1167-1174. doi: 10.1016/S1473-3099(15)00074-2. Epub 2015 Jul 16. PMID 26189433
- [Background] Yurdaydin C, et al. Optimizing the Prenylation Inhibitor Lonafarnib Using Ritonavir Boosting in Patients with Chronic Delta Hepatitis. EASL 2015, Abstract 0118.
- See also: Eiger BioPharmaceuticals, Inc. company website — http://eigerbio.com